CLINICAL TRIAL: NCT06171243
Title: Pilot Study: Measurement of Plasma Levels of Lidocaine/Tetracaine and Adverse Effects Derived From a New Topical Formulation for Treatment of Neuropathic Pain
Brief Title: PK of Lidocaine/Tetracaine and PD Derived From a New Topical Formulation for Treatment of Neuropathic Pain.
Acronym: PK/PDLido
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, María Francisca Elgueta Le-beuffe, Associated Professor, Pontificia Universidad Catolica de Chile
Other Study IDs: 210821002
Record Dates: First submitted 2023-09-21; First posted 2023-12-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Neuralgia; Neuropathic Pain; Local Anesthetic Complication; Lidocaine Adverse Reaction
Keywords: neuralgia; Neuropathic pain; Local Anesthetic; Lidocaine
MeSH Terms: conditions — Neuralgia | interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PK/PDLido: Patients over 50 years old, with neuropathic pain who are hospitalized at UC-Christus Clinical Hospital, will be candidates for recruitment to the study.
  Interventions: Drug: Lidocaine topical

INTERVENTIONS:
Drug: Lidocaine topical — Patients who agree to participate, will be given the Lidocaine 23%/Tetracaine 7% formulation. The application of the cream will be carried out by a researcher in charge:
  1. A skin area of 200 cm2 will be delimited for the application of the formulation throughout the study period.
  2. 10 grams will be applied every 12 hours for a period of 48 hours.
  Other Names: Lidocaine/Tetracaine

SUMMARY:
Post-herpetic neuralgia (PHN) is the most frequent complications related to herpes zoster, and can persist for months or even years, and require extensive treatment. For this purpose, pharmacological therapies based on tricyclic antidepressants (amitriptyline), central nervous system depressants (pregabalin) and also opioids, have been stablished. However, all the drugs mentioned can cause serious systemic adverse effects that worsen the patient's quality of life. To avoid these complications, topical therapies based on Capsaicin or Lidocaine 5% patches have been developed. However, these treatments have shown dissimilar results in controlling PHN, so a mixed formulation of lidocaine/tetracaine could show better results. For these reasons, the main objective of our work is to evaluate the plasma levels of lidocaine derived from the application of a topical formulation of lidocaine derived from the application of a topical formulation of lidocaine 23%/tetracaine 7% in patients with neuropathic pain.

DETAILED DESCRIPTION:
The International Association for the Study of Pain (IASP), defines neuropathic pain as "pain caused by injury or pathology of the somatosensory system", which is usually moderate to severe intensity, with a clinical course that can last several years, and that, therefore, can significantly affect the quality of life of the person who suffers from it. Neuropathic pain can have a central or peripheral origin. In the case of peripheric origin, conditions such as diabetic neuropathy, trigeminal neuralgia and post-herpetic neuralgia distinguish, among others. Post-herpetic neuralgia (PHN) is the most frequent complication related to Herpes Zoster, appearing in 10 to 34% of infected patients. It can persist for months, or even years, and require an extensive treatment, which can cause a huge deterioration in the quality of patients life. It is often installed as a debilitating, intense and refractory neuropathic pain to most of the strategies tried, and its treatment is usually a real challenge, since therapeutic alternatives are often exhausted, without the patient being able to obtain real pain relief. Thus, for example, after 1 year, almost 10% of patients persist with PHN, most of them being elderly and generally, fragile. Some of the risk factors described for the appearance of PHN, are the extension, severity and duration of the skin rash, age, severe immunosuppression, a concomitant autoimmune pathology, diabetes, cancer, recent physical trauma and psychological comorbidity, among others. In fragile patients, more than one risk factor is usually associated, increasing the probability of developing PHN. In individuals 85 years old or older, the risk increases to 50%.

Regarding to post-herpetic neuralgia´s pathophysiology, it has been defined that herpes zoster can affect both peripheral and central nerves, with two processes that are important in the development of pain: desensitization and deafferentation. Some studies have also shown an increase in the number of voltage-gated sodium channels, alterations in voltage-gated potassium channels, and an increase in the number of TRPV1 receptors in animal models of neuropathic pain. Other mechanisms associated with the development of PHN are related to the loss of GABAergic neurons and increased release of pro-inflammatory mediators in the damaged tissue, such as: substance P, bradykinins, histamine, cytokines and ions (H+ y K+).

Considering the pathophysiology of PHN, pharmacological therapies have been established, that aim to relieve pain since the onset of herpes zoster and prevent associated complications. Regarding the use of tricyclic antidepressants for pain management, it has been estimated that they generate a good response in the patient, but with a series of adverse effects, due to their systemic administration, such as: anticholinergic effects (dry mouth, constipation, urinary retention, nausea, blurred vision and orthostatic hypotension), arrhythmias (prolongation of the QT interval, Torsades de Pointes) and sudden death in susceptible patients. On other hand, treatments for PHN based on the administration of drugs that depress the nervous system, such as antiepileptic drugs (pregabalin and gabapentin) or opioids, can cause adverse reactions, such as drowsiness, edema, ataxia and constipation. To avoid these adverse effects, reduce pharmacological interactions and improve adherence to treatment, pharmacological alternatives have been proposed for topical administration based on Capsaicin (TRPV1 agonist) or lidocaine (local anesthetic, sodium channel blocker).

Lidocaine is one of the most widely used local anesthetics, in various presentations for topical use, to relieve or prevent pain in dermatological procedures, such as removal of tattoos and skin blemishes, management of burns, among others. In chronic pain, a systematic review that included 12 primary studies, with a total of 508 participants, compared the effectiveness of various topical formulations of lidocaine (5% cream, 5% patch, 5% gel and 8% spray) versus placebo in treating neuropathic pain. Effectiveness was observed, but in a small number of patients. The authors concluded that further studies are needed to determine efficacy and safety of these topical lidocaine preparations in the management of neuropathic pain. Another presentation of 5% lidocaine for the management of neuropathic pain was an "adhesive cream" (or plaster) format. This pharmaceutical form is applied and remains deposited on the skin for 12 hours. Only 3% of the applied lidocaine reaches the plasma, to be later metabolized in the liver, and excreted by the kidneys, with a plasma half-life of 7.6 hours. However, this 5% formulation was not very effective and its cost is very high. Formulations with a higher concentration of local anesthetic could be effective in a greater number of patients, but we do not know the pharmacokinetic behaviour that they could present in a population of elderly patients.

Subsequently, and in order to improve the analgesic effect of lidocaine, and also broaden the spectrum of use of this intervention, topical preparations have been developed, that combine lidocaine together with other local anesthetics of ester nature, such as lidocaine/prilocaine and lidocaine/tetracaine. The rationale for this combination is given by the pharmacokinetic characteristics of each compound. The anesthesia produced by lidocaine is rapid and intense. Tetracaine, being more lipophilic than lidocaine, concentrates in the stratum corneum of the epidermis, from where it diffuses slowly, its duration is longer, and its systemic uptake is limited. According to the data obtained in a clinical study with 40 patients, the combination of both anesthetics produces a fast-onset topical anesthesia, but with a mean duration of 11 hours. The systemic absorption of both local anesthetics is related to both application period and the exposed surface area. In this area, there are different studies that support the efficacy, clinical safety and patient satisfaction with the topical use of lidocaine/tetracaine used in short-term dermatological procedures. A study testing higher doses of lidocaine 23%/tetracaine 7% on the face of 52 healthy young subjects and maintained for 2 hours, showed that the plasma concentration of lidocaine remained at safe levels for each subject, and only correlated with some topical adverse reactions, such as local irritation and dermatitis. However, compounds with non-standarized doses, used over time and in excessive application area, can lead to dangerous results. Currently, there are no defined protocols that allow the safe use of mixed topical anesthetic formulations and therefore, the need to create a safe clinical profile is crucial.

Based on the information presented previously, we considerate that a topical formulation of 23% lidocaine/7% tetracaine, could be useful for the treatment of post herpetic neuropathy during chronic treatment. However, nothing has been studied about the efficacy in daily use for PHN, nor has its safety profile been evaluated in fragile patients, such as those who develop this clinical condition. For these reasons, it seems important to document, initially, the extension of the systemic absorption of lidocaine after the application of this eutectic mixture of Lidocaine/Tetracaine in patients with neuropathic pain and to correlate these levels with the appearance of adverse effects. The results of this study will allow us to obtain data that will help us prepare a subsequent clinical study, where the efficacy of our formulation will be evaluated versus a standard treatment against post-herpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Trigeminal neuralgia
* Postherpetic neuralgia
* Diabetic neuropathy
* Chronic postoperative pain
* Complex regional pain syndrome
* HIV neuropathy
* Peripheral neuropathy

Exclusion Criteria:

* Intravenous lidocaine and/or other treatment interfering with the protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Lidocaine plasmatic levels measured by high performance liquid chromatography | From first application of the cream, which will be applied every 12 hours, to 48 hours after the first application
  Lidocaine total dose, after using Lidocaine 23%/Tetracaine 7% formulation.10 grams will be applied every 12 hours for a period of 48 hours.
  Time "0", where time "0" corresponds to the moment of application of the cream for the first time.
  Group M1 (Sample N1: 30 min, N2: 2 hours, N3: 4 hours, N4: 12 hours, N5: 26 hours) Group M2 (Sample N1: 45 min, N2: 3 hours, N3: 8 hours, N4: 18 hours, N5: 32 hours) Group M3 (Sample N1: 60 min, N2: 4 hours, N3: 12 hours, N4: 24 hours, N5: 38 hours) Group M4 (Sample N1: 90 min, N2: 5 hours, N3: 16 hours, N4: 30 hours, 44 hours)

SECONDARY OUTCOMES:
Number of Participants with Blood Pressure adverse reactions | From first application of the cream, which will be applied every 12 hours, to 48 hours after the first application
  Systolic and Diastolic Blood Pressure
  Group M1 (Sample N1: 30 min, N2: 2 hours, N3: 4 hours, N4: 12 hours, N5: 26 hours) Group M2 (Sample N1: 45 min, N2: 3 hours, N3: 8 hours, N4: 18 hours, N5: 32 hours) Group M3 (Sample N1: 60 min, N2: 4 hours, N3: 12 hours, N4: 24 hours, N5: 38 hours) Group M4 (Sample N1: 90 min, N2: 5 hours, N3: 16 hours, N4: 30 hours, 44 hours)
Number of Participants with appearance of Heart rate adverse reactions | From first application of the cream, which will be applied every 12 hours, to 48 hours after the first application
  Heart rate will be measured:
  Group M1 (Sample N1: 30 min, N2: 2 hours, N3: 4 hours, N4: 12 hours, N5: 26 hours) Group M2 (Sample N1: 45 min, N2: 3 hours, N3: 8 hours, N4: 18 hours, N5: 32 hours) Group M3 (Sample N1: 60 min, N2: 4 hours, N3: 12 hours, N4: 24 hours, N5: 38 hours) Group M4 (Sample N1: 90 min, N2: 5 hours, N3: 16 hours, N4: 30 hours, 44 hours)
Number of Participants with appearance of Adverse Drug Reactions | From first application of the cream, which will be applied every 12 hours, to 48 hours after the first application
  Appearance of Adverse Drug Reactions, such as
  Group M1 (Sample N1: 30 min, N2: 2 hours, N3: 4 hours, N4: 12 hours, N5: 26 hours) Group M2 (Sample N1: 45 min, N2: 3 hours, N3: 8 hours, N4: 18 hours, N5: 32 hours) Group M3 (Sample N1: 60 min, N2: 4 hours, N3: 12 hours, N4: 24 hours, N5: 38 hours) Group M4 (Sample N1: 90 min, N2: 5 hours, N3: 16 hours, N4: 30 hours, N5: 44 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Iturra, PhD, Principal Investigator — Proffesor
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided